CLINICAL TRIAL: NCT00679978
Title: Vertebral Fracture and Osteonecrosis of the Femoral Head Associated With High-dose Glucocorticoid Therapy
Brief Title: Vertebral Fracture and Osteonecrosis Associated With High-dose Glucocorticoid
Status: Completed | Type: Observational
Sponsor: Saitama Medical University (Other)
Responsible Party: Hideto Kameda, Department of Rheumatology/Clinical Immunology, Saitama Medical Center
Other Study IDs: SaitamaVFOFH; 14211301
Record Dates: First submitted 2008-05-14; First posted 2008-05-19 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Vertebral Fracture; Osteonecrosis; Rheumatic Diseases
Keywords: osteoporosis; glucocorticoid; bone mineral density; osteonecrosis of the femoral head
MeSH Terms: conditions — Spinal Fractures; Osteonecrosis; Rheumatic Diseases; Osteoporosis; Legg-Calve-Perthes Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: A: etidronate

SUMMARY:
Osteoporotic vertebral fracture (VF) and osteonecrosis of the femoral head (OFH) are major concerns in patients with systemic rheumatic diseases treated with high-dose glucocorticoids (GCs). The investigators examined and compared the incidence and risk factors of VF with those of OFH in patients who had recently received high-dose GC therapy to clarify the relationship between these two complications.

DETAILED DESCRIPTION:
Patients with rheumatic diseases receiving GCs (≧0.5 mg/kg/day for prednisolone equivalent) within the past 2 months were enrolled in this study, and treated with 200 mg/day of etidronate cyclically. The bone mineral density (BMD) of lumbar spines (L2-4) was examined by QDR2000. OFH was evaluated by magnetic resonance imaging (MRI). ClinicalTrials.gov identifier: NCT00679978.

Forty-four patients completed the 2-year study including annual X-rays and the BMD analysis. MRI evaluation at entry and 2 years was performed in 41 patients. The BMD values with anteroposterior (AP) and lateral views decreased by 6.4% and 9.7% respectively in the first year, but were stable in the second year. Eleven patients developed VF and 9 patients developed OFH. The risk factors for VF included previous VF and a low BMD value (T score < -1.5) of AP view at baseline with odds ratio (OR) 14.9 (95%CI 2.9-76.4), while the risk factor for OFH was the recent maximum GC dosage (>1.2 mg/kg/day versus ≦; OR=7.7, 95%CI 1.3-45.5) and the decrease in BMD value of lateral view (>15% versus ≤; OR=6.7, 95% CI 1.2-36.1) in the first year.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to our hospital for the treatment of active systemic rheumatic diseases taking at least 0.5 mg/kg/day for PSL equivalent between January 2001 and June 2003 were eligible for this prospective study

Exclusion Criteria:

* Patients who were not appropriate for this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our hospital for the treatment of active systemic rheumatic diseases taking at least 0.5 mg/kg/day for PSL equivalent
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2001-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
new vertebral fracture | 2 years

SECONDARY OUTCOMES:
osteonecrosis of the femoral head | 2 years

REFERENCES:
- [Result] Kameda H, Amano K, Nagasawa H, Ogawa H, Sekiguchi N, Takei H, Suzuki K, Takeuchi T. Notable difference between the development of vertebral fracture and osteonecrosis of the femoral head in patients treated with high-dose glucocorticoids for systemic rheumatic diseases. Intern Med. 2009;48(22):1931-8. doi: 10.2169/internalmedicine.48.2414. Epub 2009 Nov 16. PMID 19915292